CLINICAL TRIAL: NCT04054609
Title: Evaluation Of Prognostic Value of 18f-Fluoroazomycin Arabinoside (FAZA) Positron Emission Tomography/Magnetic Resonance Imaging (PET/MR) In Patients With Critical Limb Ischemia Pre- and Post Revascularization: a Pilot Study
Brief Title: FAZA PET/MRI in CLI Patients Pre and Post Revascularization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-6114
Record Dates: First submitted 2019-08-01; First posted 2019-08-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: FAZA PET/MRI scan pre and post standard of care endovascular treatment for critical limb ischemia patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAZA PET/MRI scan (Other): PET/MRI scan using radiotracer 18F-Fluoroazomycin Arabinoside
  Interventions: Diagnostic Test: FAZA PET/MRI scan

INTERVENTIONS:
Diagnostic Test: FAZA PET/MRI scan — PET/MRI scan using radio tracer named 18F-Fluoroazomycin Arabinoside (FAZA) pre and post standard of care endovascular treatment for critical limb ischemia patients

SUMMARY:
Peripheral artery disease is a worldwide problem, leading to high mortality and mobility.

Critical limb ischemia (CLI) is associated with high risk of amputation with the subsequent decreased in life quality. Endovascular therapy is now considered the primary treatment option in these patients to improve the vascularity and prevent amputations.

In recent years, development of molecular imaging tools are now become available. A recent radio tracer named 18F-Fluoroazomycin Arabinoside (FAZA) its an specific marker of hypoxia in the tissues and has been used in multiples studies. This tracer can be used in PET/MR scan providing a potentially power diagnostic tool in patients with CLI, allowing in one diagnostic study the evaluation of location and degree of hypoxia in the extremity tissues. This diagnostic tool may offer a better assessment pre and post standard of care endovascular treatment for the patients.

Moreover, some of the patients treated with endovascular therapy may not have a favorable outcome, without a clear reason explaining this situation. We will try to find some predictor model in the FAZA PET/MR that can explain the different outcomes and may help clinicians choose the best treatment option in specific cases.

Thirdly, post processing for optimization of the MR sequences in patients with CLI will be performed at the MR component of the PET. There would thus be great clinical interest in developing non-invasive tools that could provide more accurate diagnostic information compared to traditional tests for these patients population.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years;
* Patients with clinical evidence of critical limb ischemia that are candidates for revascularization treatment;
* A negative urine or serum pregnancy test in women of child-bearing age;
* Ability to provide written informed consent to participate in the study.

Exclusion Criteria:

* Contraindication for MR as per current institutional guidelines;
* Inability to lie supine for at least 30 minutes;
* Pregnant or breastfeeding;
* Unable or unwilling to provide informed consent;
* Impending amputation within 6 weeks of presentation;
* Previous metallic hardware in the lower limbs;
* Unable to have ethanol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Validation of FAZA PET/MRI as a biomarker of hypoxia | FAZA PET/MRI 2-3 weeks before endovascular treatment and 4-6 weeks after endovascular treatment
  The change of degree and pattern of 18F-Fluoroazomycin Arabinoside (FAZA) uptake in the PET/MRI scan of limb in patients with critical limb ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Veit-Haibach, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Farag A, Kohan A, Sekine T, Mirshahvalad SA, Metser U, Mafeld S, Tan K, Veit-Haibach P. Measuring hypoxia in chronic limb-threatening ischemia using 18F-FAZA kinetic modelling - a pilot study. EJNMMI Res. 2025 Apr 26;15(1):48. doi: 10.1186/s13550-025-01243-5. PMID 40287606